CLINICAL TRIAL: NCT04089982
Title: Pilot Study on Varenicline in Light and Intermittent Smokers
Brief Title: Varenicline Light Smoking Pilot
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00103506
Record Dates: First submitted 2019-09-12; First posted 2019-09-16 (Actual); Results first posted 2021-05-11 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Smoking Cessation; Smoking Behaviors; Smoking
MeSH Terms: conditions — Smoking Cessation; Smoking | interventions — Varenicline

STUDY DESIGN:
Intervention Model Description: 2-arm randomized, placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Varenicline (Active Comparator): Varenicline BID
  Interventions: Drug: Varenicline
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Varenicline — Chantix
  Arms: Varenicline
Drug: Placebo oral tablet — Placebo
  Arms: Placebo

SUMMARY:
The goal of this study is to assess varenicline vs. placebo for its effect on decreasing cue reactivity in light and intermittent smokers.

DETAILED DESCRIPTION:
The study will consist of randomization to receive either varenicline or placebo over 6 weeks and include 5 study visits. Participants are offered an optional additional 6 weeks of active varenicline. Cue reactivity will be assessed in both a lab-based setting (viewing series of images and rating cravings) and in a real-world setting (text-based daily interaction).

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or above
2. Daily smoker using 10 or less cigarettes per day but a minimum of at least 1 cigarettes per week or 4 cigs/month.
3. Must be able to make it through a 24-hour period without nicotine withdrawal symptoms (specifically does not have new onset of irritability, headaches, insomnia, or intense cravings).
4. Willing to quit smoking in the next 30 days
5. Is able to provide written informed consent (in English) to participate in the study and is able to read/understand the procedures and study requirements.
6. Is willing to voluntarily sign and date an informed consent form that is approved by an institutional review board before the conduct of any study procedure.
7. If female and of childbearing potential, is willing to use medically acceptable contraceptive measures for the duration of the study. Acceptable methods of contraception include (1) surgical sterilization (such as tubal ligation or hysterectomy, (2) approved hormonal contraceptives (such as birth control pills, patches, implants or injections), (3) barrier methods (such as condom or diaphragm) used with a spermicide, or (4) an intrauterine device (IUD). Contraceptive measures such as rhythm method or Plan B™, sold for emergency use after unprotected sex, are not acceptable methods for routine use.
8. Have access to a cell phone that can send and receive SMS text messages.

Exclusion Criteria:

1. Use of a smoking cessation medication (e.g. nicotine replacement, varenicline, bupropion) in last 30 days.
2. Current use of tobacco product other than cigarettes (e.g. e-cigarettes, smokeless tobacco) in the last 30 days
3. Answer > 0 on suicidality question of Patient Health Questionnaire (PHQ-9) Depression Scale
4. Active alcohol use disorder or hazardous drinking. This will be screened with the AUDIT-C, and positive scores (4 or greater for men and 3 or greater for women)54,55 will result in study clinician assessment and discretion.
5. Use of illicit drugs in the last month (marijuana, cocaine, opiates, benzodiazepines, and/or methamphetamine)
6. Severe symptomatic depression and or anxiety (study medical provider discretion)
7. Diagnosis of bipolar disorder, schizophrenia, PTSD and or adult ADHD (study medical provider discretion)
8. Chronic medical illness including diabetes with the use of insulin, Hemoglobin A1c > 7 (study medical provider discretion), heart disease diagnosed by angiogram, or COPD diagnosed by pulmonary function testing and requiring an oxygen supply
9. Specific medications (Appendix 1)
10. Abnormal finding on physical exam (study medical provider discretion)
11. Positive Urine Pregnancy Test (women of child bearing potential only; QuickVue Urine Pregnancy)56
12. Positive Urine Toxicology-5 Screen (methamphetamine, cocaine, opiates, benzodiazepines, THC)
13. Unstable hypertension (Blood pressure > 160/100)
14. Renal failure with active or pending hemodialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Davis, MD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Varenicline | Placebo
Started | 6 | 5
Completed | 6 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Varenicline | Placebo | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.8 (7.1) | 42.6 (12.7) | 38.4 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 4 | 1 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 5 | 5 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 0 | 1 | 1
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Change in Self-Reported Craving Level Via Lab-Based Cue Reactivity
Description: Participants were asked to self-report craving level to smoke on a scale of 1-10 with 1 corresponding to no craving and 10 corresponding to intense craving. Self-reported craving level was requested following presentation of multiple images on a screen over a 20 minute period. Four types of images were presented - neutral affect, negative affect, smoking and social images.
Time Frame: Baseline, Visit 4 (week 6)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 6 | 5
score on a scale
  Baseline | 6.31 (2.80) | 4.2 (1.8)
  Week 6 | 2.56 (2.11) | 2.4 (1.3)

2. Secondary Outcome: Change in Self-Reported Craving Level Via Real-World Cue Reactivity
Description: Craving level in "real world" situations was assessed through electronic momentary assessment (EMA). Participants were instructed to send a text to the study team each time they experienced craving to smoke a cigarette. Self-report craving level to smoke was reported on a scale of 1-10 with 1 corresponding to no craving and 10 corresponding to intense craving.
Time Frame: Baseline, Visit 4 (week 6)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 6 | 5
score on a scale
  Baseline | 7.15 (1.1) | 6.7 (1.8)
  Week 6 | 5.5 (0.5) | 8 (0)

3. Secondary Outcome: Changes in Smoking
Description: 7-day point prevalence smoking abstinence. This will be measured through self-reported daily smoking diaries and daily text messaging.
Time Frame: Screening visit, Visit 4 (week 6)
Measure: Mean (Standard Deviation); unit: cigarettes per day
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 6 | 5
cigarettes per day
  Baseline | 3.6 (3.4) | 5.2 (2.3)
  Week 6 | 0.5 (0.8) | 2.6 (3.2)

4. Secondary Outcome: Medication Adherence
Description: Medication adherence is measured by composite self-reported diaries and daily text messaging responses.
Time Frame: Screening visit, Visit 4 (week 6)
Measure: Mean (Standard Deviation); unit: Percent medication adherence
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 6 | 5
Percent medication adherence | 91.6 (0.08) | 90.3 (0.13)

5. Secondary Outcome: Medication Tolerance by Self-Reported Side Effects
Description: Self-reported side effects (open ended survey questions) with a ranking scale of 1-2 (mild), 3-5 (moderate), and 6-7 (severe). Any side effect 3 or greater will be reviewed by a study medical provider.
Time Frame: Up to 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 6 | 5
Participants
  Abnormal/Vivid Dreams | 1 | 2
  Nausea/Vomiting | 1 | 1
  Constipation | 1 | 0
  Dizziness/Lightheadedness | 1 | 0
  Dry Mouth | 1 | 0
  Fatigue | 0 | 2
  Insomnia/Trouble Sleeping | 0 | 1

6. Secondary Outcome: Changes in Smoking Abstinence
Description: 7-day point prevalence smoking abstinence confirmed by CO <7ppm. This will be measured through biochemical confirmation (CO breath test).
Time Frame: Screening visit, Visit 4 (week 6)
Measure: Mean (Standard Deviation); unit: ppm
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 6 | 5
ppm
  Baseline | 9.5 (11.1) | 10.2 (3.7)
  Week 6 | 2.6 (1.5) | 7.8 (5.5)

ADVERSE EVENTS:
Time Frame: Up to 12 weeks
Arm/Group | Varenicline | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/5
Serious Adverse Events (participants affected / at risk) | 1/6 | 0/5
Other Adverse Events (participants affected / at risk) | 5/6 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Varenicline (N=6) | Placebo (N=5)
Asthma flare (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Varenicline (N=6) | Placebo (N=5)
Abnormal/Vivid Dreams (Psychiatric disorders) | 1 | 2
Nausea/Vomiting (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Dizziness/Lightheadedness (General disorders) | 1 | 0
Dry Mouth (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 0 | 2
Insomnia/Trouble Sleeping (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-03): https://cdn.clinicaltrials.gov/large-docs/82/NCT04089982/Prot_SAP_000.pdf